CLINICAL TRIAL: NCT03225079
Title: PERFORM = Pentaglobin® Registry For Outcome Report and Monitoring, International Registry on the Use of Pentaglobin® in Patients With Severe Bacterial Infections
Brief Title: PERFORM = Pentaglobin® Registry For Outcome Report and Monitoring
Acronym: PERFORM
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZKSJ0103_PERFORM
Record Dates: First submitted 2017-06-27; First posted 2017-07-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Severe Bacterial Infection
Keywords: Pentaglobin® use; severe bacterial infection
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
International registry on the use of Pentaglobin® in patients with severe bacterial infections; multicentric, international registry, non-interventional trial

DETAILED DESCRIPTION:
Aim of the Pentaglobin® registry of adult critically ill patients with severe infections is primarily to assess the effects of IVIgAM on the aforementioned outcome parameters and its side effects under real-life conditions based on a prospective, high-quality data documentation

* Age ≥ 18 years
* Diagnosis of severe bacterial infection
* Pentaglobin® use
* signed informed consent for data collection

Exclusion criteria None

Primary endpoints

* Comparison APACHE II and SAPS II predicted mortality vs. observed hospital mortality and
* Difference in SOFA scores, baseline vs. posttreatment (24 h after last application) assessment

Secondary endpoints

* In-hospital mortality total and in subgroups according to baseline IgM serum levels (< 80 mg/dL vs. ≥ 80 mg/dL) and baseline CRP (< 70 mg/L vs. ≥ 70 mg/L)
* Change in MOF score from the day before treatment start till 24 h after last application of Pentaglobin
* Course of laboratory markers (concentration-difference): CRP, procalcitonin, IL-6, IgM, IgA, IgG before treatment start till 24 h after last application as far as available in the centers
* Duration of ICU stay (days)
* Duration of hospital stay (days)
* Time from onset of severe bacterial infection to start of treatment

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Diagnosis of severe bacterial infection
* Pentaglobin® use
* signed informed consent for data collection -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will be primarily based on a severe bacterial infection of a patient and the following application of Pentaglobin®.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
APACHE II and SAPS II predicted mortality vs. observed hospital mortality and | up to 6 months
  predicted mortality vs. observed hospital mortality
difference in SOFA scores, baseline vs. posttreatment (24 hours after last application) assessment | baseline and 24 hours after last application of Pentaglobin
  change in SOFA scores, baseline vs. posttreatment (24 hours after last application)

SECONDARY OUTCOMES:
In-hospital mortality total and in subgroups according to baseline IgM serum levels and baseline CRP | up to 6 months
  In-hospital mortality total and in subgroups according to baseline IgM serum levels and baseline CRP
Change in MOF score from the day before treatment start till 24 hours after last application of Pentaglobin | period between baseline and 24 hours after last application of Pentaglobin
  Change in MOF score from the day before treatment start till 24 hours after last application of Pentaglobin
Course of laboratory markers (concentration-difference): CRP, procalcitonin, IL-6, IgM, IgA, IgG before treatment start till 24 h after last application as far as available in the centers | period between baseline and 24 hours after last application of Pentaglobin
  IL-6, IgM, IgA, IgG before treatment start till 24 hours after last application as far as available in the centers
Duration of ICU stay (days) | up to 6 months
  Duration of ICU stay (days)
Duration of hospital stay (days) | up to one year
  Duration of hospital stay (days)
Time from onset of severe bacterial infection to start of treatment | up to 14 days
  Time from onset of severe bacterial infection to start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Brunkhorst, Prof.Dr., Study Director — Jena University Hospital, Center for Clinical Studies
Locations (12):
- Hospital Sirio Libanes, São Paulo, Brazil
- Hospital Universitario Erasmo Meoz, Cúcuta, Colombia
- Germany (8):
  - Clinic for Neurology, Jena, Thuringia
  - Erzgebirgsklinikum Annaberg, Annaberg
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Knappschaftskrankenhaus, Bochum
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikums Gießen & Marburg (UKGM), Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Tübingen, Tübingen
- Turkey (Türkiye) (2):
  - Atatürk University Medical Faculty Trainer Hospital, Erzurum
  - Eskişehir Osmangazi üniversitesi tıp fakültesi hastanesi, Eskişehir

IPD SHARING:
Plan to Share IPD: No